CLINICAL TRIAL: NCT01885182
Title: A Phase III, Randomized, Double-blind, Double-dummy, Parallel Group Study to Determine the Safety and Efficacy of Oxy/Nal Prolonged Release Tablets Compared to Oxy PR in Subjects With Moderate to Severe, Chronic Cancer Pain
Brief Title: Determine the Safety and Efficacy of Oxy/Nal Tablets Compared to Oxy PR in Subjects With Cancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma (China) Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OXN10-CN-303
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-05

CONDITIONS: Cancer; Pain
MeSH Terms: conditions — Neoplasms; Pain | interventions — Oxycodone; Naloxone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxycodone/Naloxone (Experimental): 5/2.5mg, 10/5mg, 20/10mg or 40/20mg
  Interventions: Drug: Oxycodone/Naloxone
- Oxycodone (Active Comparator): 5mg, 10mg, 20mg or 40mg
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone/Naloxone
  Other Names: Targin
  Arms: Oxycodone/Naloxone
Drug: Oxycodone
  Other Names: OXY PR
  Arms: Oxycodone

SUMMARY:
To Determine the Safety and Efficacy of Oxycodone / Naloxone Prolonged Release Tablets compared to Oxycodone PR in Subjects with Moderate to Severe, Chronic Cancer Pain

DETAILED DESCRIPTION:
This is a randomised, double-blind, double-dummy, parallel group study using OXN and OXY PR to treat moderate to severe, chronic cancer pain. Subjects with documented history of cancer pain that requires around the clock opioid therapy will be included. Subjects must have a medical history of constipation that was induced by, or worsened by their opioid therapy.

ELIGIBILITY:
Inclusion Criteria

Males & females, at least 18 years or older with a diagnosis of cancer.

Females less than one year post-menopausal must have a negative urine pregnancy test recorded prior to the first dose of study medication, be non-lactating, & willing to use adequate & highly effective method of contraception throughout the study. Highly effective methods of birth control are defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently correctly such as sterilisation, implants, injectables, combined oral contraceptives, some IUDs (hormonal), sexual abstinence or vasectomised partner.

Subjects who are receiving WHO step II or Step III analgesic medication who have constipation induced, or worsened by their opioid medication, as shown by

1. the subject's medical need of regular intake of laxatives to have at least 3 bowel evacuations per week, or having less than 3 bowel evacuations when not taking a laxative, respectively.
2. the subject's self-assessment that their constipation was induced or worsened by their current pre-study opioid medication.

Documented history of moderate to severe, chronic cancer pain that requires around the-clock opioid therapy (starting dose of oxycodone PR between 20-80 mg/day) & are likely to benefit from WHO step III opioid therapy for the duration of the study. Subjects must be willing to discontinue their current opioid analgesic routine.

Opioid medication continue at a stable or nearly stable dose in the investigator's opinion during the treatment.

Subjects are willing to discontinue pre study laxative medication & take study specific laxative medication.

Subjects taking daily fibre supplementation or bulking agents are eligible if they can be maintained on a stable dose & regimen throughout the study, & in the investigators opinion are willing & able to maintain adequate hydration.

Subjects willing & able (e.g. mental & physical condition) to participate in all aspects of the study, including use of medication, completion of subjective evaluations, attending scheduled clinic visits, completing telephone contacts, & compliance with protocol requirements as evidenced by providing written, informed consent.

Subjects already taking non-opioid analgesics & all other concomitant medications (including those for the treatment of depression) are eligible to take part in the study. However, all concomitant medications that are considered necessary for the subject's welfare should be continued at a stable dose throughout the double-blind phase of the study & under the supervision of the investigator.

Expected survival time > 3 months.

With capability of reading, understanding & signing inform consent form & compliance with protocol requirements.

Exclusion Criteria Subjects that require a dose >80 mg/day oxycodone PR at the start of the double-blind phase.

Any history of hypersensitivity to oxycodone, naloxone, morphine, bisacodyl, related products & other ingredients.

Subjects with any situation in which opioids are contra-indicated, severe respiratory depression with hypoxia & or hypercapnia, severe chronic obstructive pulmonary disease, cor pulmonal, severe bronchial asthma, paralytic ileus.

Subjects with evidence of clinically significant gastrointestinal disease (e.g. paralytic ileus, peritoneal carcinosis), significant structural abnormalities of the gastrointestinal tract (e.g. scarring, obstruction etc) either related or not related to the underlying cancer or disease progression.

Evidence of clinically significant cardiovascular, renal, hepatic or psychiatric disease, as determined by medical history, clinical laboratory tests, ECG results & physical examination, that would place the subject at risk upon exposure to the study medication or that may confound the analysis & or interpretation of the study results.

Abnormal aspartate aminotransferase (AST; SGOT), alanine aminotransferase (ALT; SGPT), r-glutamyltransferase (GGT) or alkaline phosphatase levels (>3 times the upper limit of normal) or an abnormal total bilirubin & or creatinine level(s) (greater than 1.5 times the upper limit of normal).

Cyclic chemotherapy in the two weeks before the screening visit or planned during the core study that has shown in the past to influence bowel function. If subjects are having their first cycle of chemotherapy during the 2 weeks before the screening visit or during the double-blind phase of the study they should be excluded from the study.

Radiotherapy that, in the investigators opinion, would influence bowel function or pain during the double-blind phase of the study.

Subjects with known or suspected unstable brain metastases or spinal cord compression that may require changes in steroid treatment throughout the duration of the study.

Subjects with uncontrolled seizures.

Subjects with increased intracranial pressure.

In the investigator's opinion, subjects who are receiving hypnotics or other central nervous system (CNS) depressants that may pose a risk of additional CNS depression with opioid study medication.

Subjects with myxoedema, not adequately treated hypothyroidism or Addisons disease.

Subjects who have a confirmed diagnosis of ongoing irritable bowel syndrome(IBS).

Surgery completed within 4 weeks prior to the start of the Screening Period, or planned surgery during the study that would influence pain or bowel function during the study or preclude completion of the study.

Subjects receiving opioid substitution therapy for opioid addiction (e.g. methadone or buprenorphine).

Active alcohol or drug abuse & or history of opioid abuse.

Subjects suffering from diarrhoea & or opioid withdrawal.

Subjects presently taking, or who have taken, naloxone ≤30 days prior to the start of the Screening Period.

Subjects who participated in a clinical research study involving a new chemical entity or an experimental drug within 30 days of study entry (defined as the start of the Screening Period), unless the subject is on data collection phase for Overall Survival.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2015-08-30 (Actual); Study Completion 2015-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Yu, Study Director — Mundipharma, China
Locations (28):
- China (28):
  - Fuzhou General Hospital of Nanjing Military Command of PLA, Fuzhou, Fujian
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun yat-sen univercity cancer center, Guangzhou, Guangdong
  - Hebei Medical University Fouth Hospital, Shijiazhuang, Hebei
  - Harbin Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Hubei Cancer Hospital, Changsha, Hubei
  - Tongji Hospital Tongji Medical College of HUST, Wuhan, Hubei
  - Jiangsu Cancer hospital, Nanjing, Jiangsu
  - The second hospital of Nanjing Medical university, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The second affiliated hospital of Dalian Medical university, Dalian, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The central Hospital of Jinan, Jinan, Shandong
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Tangdu Hospital,Fourth Military Medical University, Xi’an, Shanxi
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Beijing Hospital, Beijing
  - 307th hospital of Chinese People's medical sciences, Beijing
  - Beijing Cancer Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - General Hospital of Beijing Military, Beijing
  - Pejing Union Medical College Hospital, Beijing
  - Beijing Friendship Hospital, Beijing
  - The first people's hospital of shanghai, Shanghai
  - The sixth hospital of shanghai, Shanghai
  - Tianjin Cancer Hospital, Tianjin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period is from 2013 Jun to 2014 Jul and the type of location is medical clinic.
Pre-assignment Details: There is no run-in period for this study.
Groups:
- Oxycodone/Naloxone: 5/2.5mg, 10/5mg, 20/10mg or 40/20mg
  Oxycodone/Naloxone
- Oxycodone: 5mg, 10mg, 20mg or 40mg
  Oxycodone
Period: Overall Study
Arm/Group | Oxycodone/Naloxone | Oxycodone
Started | 117 | 115
Safety Population | 114 | 111
FAP Population | 107 | 106
Completed | 83 | 93
Not Completed | 34 | 22
Not completed — Adverse Event | 11 | 13
Not completed — Withdrawal by Subject | 13 | 6
Not completed — Lost to Follow-up | 2 | 2
Not completed — Lack of Efficacy | 8 | 1

BASELINE CHARACTERISTICS:
Population: FAP population
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxycodone/Naloxone | Oxycodone | Total
Number analyzed (Participants) | 107 | 106 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (11.5) | 60.0 (11.8) | 58.8 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 45 | 97
  Male | 55 | 61 | 116
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 107 | 106 | 213
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — Population: one patient data was missing
  kg/m2
    number analyzed (Participants) | 107 | 105 | 212
    (all) | 21.9 (3.5) | 21.7 (3.4) | 21.8 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: The Change of BFI-Bowel Function Index at visit8
Description: BFI is the mean of NAS for the following items:
  * Ease of defecation
  * Feeling of incomplete bowel evacuation.
  * Personal judgment of constipation. NAS was a measure of 0-100 where 0 was easy/no difficulty/not at all and 100 was severe difficulty/very strong,total score range is 0-300.Do higher values represent a worse outcome.
Time Frame: Visit8, visit8 taking place at week 4 or after early discontinuation/withdrawal from study
Population: below presents the mean BFI at final visit, primary analysis in FAP.
Measure: Mean (Standard Deviation); unit: score on BFI
Arm/Group | Oxycodone/Naloxone | Oxycodone
Number analyzed (Participants) | 107 | 106
score on BFI | 48.3 (25.7) | 51.2 (26.4)

2. Primary Outcome: The Change of BPI-SF at visit8
Description: Brief pain inventory short-form(BPI-SF) recorded at final visit assesses subject's average pain over the last 24 hours. score range is 0(no pain)-10(pain as bad as you can imagine).Do higher values represent a worse outcome.
Time Frame: Visit8, visit8 taking place at week 4 or after early discontinuation/withdrawal from study
Population: FAP
Measure: Mean (Standard Deviation); unit: Score on BPI-Brief Pain Index
Arm/Group | Oxycodone/Naloxone | Oxycodone
Number analyzed (Participants) | 107 | 106
Score on BPI-Brief Pain Index | 3.7 (1.7) | 3.6 (2.0)

3. Secondary Outcome: The Change of Symptoms of Constipation Based on Laxative Use From visit5 to visit8
Description: At Visit 5(day7) and visit8(day28) number of bisacodyl taken(Number of laxative tablets took during the last 7 days (per week) and Daily number of laxative tablets took during the last 7 days (per day)*) for OXN PR and OXY PR groups.
Time Frame: visit 5 (week 1) to visit8 (week 4 or early discontinue/withdrawal from study)
Population: FAP
Measure: Mean (Standard Deviation); unit: laxatives/week
Arm/Group | Oxycodone/Naloxone | Oxycodone
Number analyzed (Participants) | 107 | 106
laxatives/week
  Weekly number of bisacodyl taken at Visit5 | 2.1 (2.6) | 2.5 (2.6)
  Weekly number of bisacodyl taken at Visit8 | 2.2 (2.9) | 2.2 (2.8)

4. Secondary Outcome: The Change of Rescue Medication Use From visit5 to visit8
Description: The average daily dose of rescue medication (Morphine Sulfate Tablet) for OXN PR group and OXY PR group at Visit 5(first week of double blind) and at Visit 8(last week of double blind).
Time Frame: visit 5 (week 1) to visit8 (week 4 or early discontinue/withdrawal from study)
Population: FAP
Measure: Mean (Standard Deviation); unit: Morphine Sulfate mg/day
Arm/Group | Oxycodone/Naloxone | Oxycodone
Number analyzed (Participants) | 107 | 106
Morphine Sulfate mg/day
  V5: number analyzed (Participants) | 106 | 103
  V5 | 18.5 (21.4) | 13.9 (18.9)
  V8: number analyzed (Participants) | 83 | 93
  V8 | 15.4 (22.1) | 15.5 (20.1)

5. Secondary Outcome: The Change of Modified Subjective Opiate Withdrawal Scale (SOWS) From Visit1 to visit3,visit1 to visit9
Description: to compare the Modified SOWS's Change from Visit 1(day-10-0) to Visit 3(day1),Change from Visit 1 to Visit 9(day35).The SOWS was scored as the total of the 15 symptoms. each symptoms score is 0(not at all)-4(extremely).total score range is 0-60.Do higher values represent a better outcome.
Time Frame: Visit1(screening visit) to visit3 (day 1), visit1(screening visit) to visit9 (week 5)
Population: FAP
Measure: Mean (Standard Deviation); unit: score on SOWS
Arm/Group | Oxycodone/Naloxone | Oxycodone
Number analyzed (Participants) | 107 | 106
score on SOWS
  Change from Visit 1 to Visit 3 | -1.2 (3.5) | -1.6 (4.6)
  Change from Visit 1 to Visit 9: number analyzed (Participants) | 96 | 100
  Change from Visit 1 to Visit 9 | -1.3 (4.8) | -1.7 (5.5)

6. Secondary Outcome: To Assess Quality of Life Based on EQ-5D
Description: To assess quality of life based on EQ-5D by subjects evaluation via patient dairy.the quality of life based on EQ-5D at Visit1 (day-10-0) and end of treatment Visit8(day28). The scarc range is 0(the best state you can imagine)-100(the worst state you can imagine).Do higher values represent a worse outcome.
Time Frame: Visit1(screening visit) to Visit8 (week 4 or after early discontinuation/withdrawal from study)
Population: FAP
Measure: Mean (Standard Deviation); unit: Score on EQ-5D
Arm/Group | Oxycodone/Naloxone | Oxycodone
Number analyzed (Participants) | 107 | 106
Score on EQ-5D
  V1 | 58.6 (17.0) | 54.4 (16.6)
  V8: number analyzed (Participants) | 94 | 100
  V8 | 59.0 (19.3) | 53.9 (20.5)

7. Secondary Outcome: The Change of Individual Items in BPI-SF(Except for Pain in Average) by Visit
Description: To compare the change of Brief pain inventory short-form (BPI-SF) 11 indivial items (except for pain in average) at visit2(day0) ,visit5(day7),visit6(day14),visit7(day21), visit8(day28). each item range (except for how much relief from treatment /medication last 24hours is 0-100%,do higher values represent a better outcome.) is 0-10, do higher values represent a worse outcome.
Time Frame: visit2 (day 0) to visit8 (week 4 or early discontinue/withdrawal from study)
Population: FAP
Measure: Mean (Standard Deviation); unit: score on BPI-SF
Arm/Group | Oxycodone/Naloxone | Oxycodone
Number analyzed (Participants) | 107 | 106
score on BPI-SF
  Rate your pain at its worst last 24hrs-V2 | 5.9 (2.1) | 6.3 (2.1)
  Rate your pain at its worst last 24hrs-V5: number analyzed (Participants) | 101 | 102
  Rate your pain at its worst last 24hrs-V5 | 5.4 (2.3) | 5.3 (2.3)
  Rate your pain at its worst last 24hrs-V6: number analyzed (Participants) | 95 | 99
  Rate your pain at its worst last 24hrs-V6 | 5.3 (2.3) | 5.2 (2.4)
  Rate your pain at its worst last 24hrs-V7: number analyzed (Participants) | 88 | 96
  Rate your pain at its worst last 24hrs-V7 | 5.0 (2.1) | 5.0 (2.3)
  Rate your pain at its worst last 24hrs-V8: number analyzed (Participants) | 94 | 100
  Rate your pain at its worst last 24hrs-V8 | 5.4 (2.2) | 5.2 (2.6)
  Rate your pain at its least last 24hrs-V2 | 2.0 (1.5) | 2.1 (1.4)
  Rate your pain at its least last 24hrs-V5: number analyzed (Participants) | 101 | 102
  Rate your pain at its least last 24hrs-V5 | 3.4 (2.2) | 3.5 (1.9)
  Rate your pain at its least last 24hrs-V6: number analyzed (Participants) | 95 | 99
  Rate your pain at its least last 24hrs-V6 | 1.9 (1.5) | 1.9 (1.6)
  Rate your pain at its least last 24hrs-V7: number analyzed (Participants) | 88 | 96
  Rate your pain at its least last 24hrs-V7 | 2.1 (1.6) | 2.1 (1.7)
  Rate your pain at its least last 24hrs-V8: number analyzed (Participants) | 94 | 100
  Rate your pain at its least last 24hrs-V8 | 2.0 (1.6) | 2.2 (1.7)
  Rate how much pain you have right now-visit2 | 3.4 (2.2) | 3.5 (1.9)
  Rate how much pain you have right now-visit5: number analyzed (Participants) | 101 | 102
  Rate how much pain you have right now-visit5 | 3.3 (2.0) | 3.3 (1.9)
  Rate how much pain you have right now-visit6: number analyzed (Participants) | 95 | 99
  Rate how much pain you have right now-visit6 | 3.1 (2.1) | 3.0 (1.9)
  Rate how much pain you have right now-visit7: number analyzed (Participants) | 88 | 96
  Rate how much pain you have right now-visit7 | 3.2 (1.9) | 3.1 (2.1)
  Rate how much pain you have right now-visit8: number analyzed (Participants) | 94 | 100
  Rate how much pain you have right now-visit8 | 3.2 (2.0) | 3.3 (2.1)
  How much relief from TRT/MED last 24hrs-visit2 | 67.3 (22.7) | 66.9 (19.0)
  How much relief from TRT/MED last 24hrs-visit5: number analyzed (Participants) | 101 | 102
  How much relief from TRT/MED last 24hrs-visit5 | 67.7 (21.4) | 67.1 (21.7)
  How much relief from TRT/MED last 24hrs-visit6: number analyzed (Participants) | 95 | 99
  How much relief from TRT/MED last 24hrs-visit6 | 67.6 (22.5) | 66.6 (21.9)
  How much relief from TRT/MED last 24hrs-visit7: number analyzed (Participants) | 88 | 96
  How much relief from TRT/MED last 24hrs-visit7 | 64.1 (23.9) | 65.8 (21.9)
  How much relief from TRT/MED last 24hrs-visit8: number analyzed (Participants) | 94 | 100
  How much relief from TRT/MED last 24hrs-visit8 | 64.7 (23.6) | 64.7 (24.2)
  Pain affect general activity last 24hrs-visit2 | 5.6 (2.5) | 5.7 (2.6)
  Pain affect general activity last 24hrs-visit5: number analyzed (Participants) | 101 | 102
  Pain affect general activity last 24hrs-visit5 | 4.6 (2.5) | 4.9 (2.6)
  Pain affect general activity last 24hrs-visit6: number analyzed (Participants) | 95 | 99
  Pain affect general activity last 24hrs-visit6 | 4.4 (2.6) | 4.9 (2.6)
  Pain affect general activity last 24hrs-visit7: number analyzed (Participants) | 88 | 96
  Pain affect general activity last 24hrs-visit7 | 4.4 (2.6) | 4.8 (2.6)
  Pain affect general activity last 24hrs-visit8: number analyzed (Participants) | 94 | 100
  Pain affect general activity last 24hrs-visit8 | 4.6 (2.6) | 5.0 (2.9)
  Pain affect mood last 24hrs-visit2 | 5.1 (2.7) | 5.6 (2.7)
  Pain affect mood last 24hrs-visit5: number analyzed (Participants) | 101 | 102
  Pain affect mood last 24hrs-visit5 | 4.6 (2.5) | 4.9 (2.6)
  Pain affect mood last 24hrs-visit6: number analyzed (Participants) | 95 | 99
  Pain affect mood last 24hrs-visit6 | 4.1 (2.5) | 4.5 (2.6)
  Pain affect mood last 24hrs-visit7: number analyzed (Participants) | 88 | 96
  Pain affect mood last 24hrs-visit7 | 3.8 (2.6) | 4.5 (2.7)
  Pain affect mood last 24hrs-visit8: number analyzed (Participants) | 94 | 100
  Pain affect mood last 24hrs-visit8 | 4.3 (2.5) | 4.5 (2.8)
  Pain affect walking ability last 24hrs-visit2 | 4.3 (2.9) | 4.7 (3.0)
  Pain affect walking ability last 24hrs-visit5: number analyzed (Participants) | 101 | 102
  Pain affect walking ability last 24hrs-visit5 | 4.0 (3.0) | 4.1 (2.9)
  Pain affect walking ability last 24hrs-visit6: number analyzed (Participants) | 95 | 99
  Pain affect walking ability last 24hrs-visit6 | 3.6 (2.8) | 4.3 (3.0)
  Pain affect walking ability last 24hrs-visit7: number analyzed (Participants) | 88 | 96
  Pain affect walking ability last 24hrs-visit7 | 3.8 (2.8) | 4.4 (3.0)
  Pain affect walking ability last 24hrs-visit8: number analyzed (Participants) | 94 | 100
  Pain affect walking ability last 24hrs-visit8 | 4.1 (2.9) | 4.6 (3.0)
  Pain affect normal work last 24hrs-visit2 | 6.3 (3.1) | 6.5 (3.2)
  Pain affect normal work last 24hrs-visit5: number analyzed (Participants) | 101 | 102
  Pain affect normal work last 24hrs-visit5 | 5.6 (3.1) | 5.4 (2.9)
  Pain affect normal work last 24hrs-visit6: number analyzed (Participants) | 95 | 99
  Pain affect normal work last 24hrs-visit6 | 5.1 (3.1) | 5.6 (3.1)
  Pain affect normal work last 24hrs-visit7: number analyzed (Participants) | 88 | 96
  Pain affect normal work last 24hrs-visit7 | 4.7 (3.0) | 5.4 (3.0)
  Pain affect normal work last 24hrs-visit8: number analyzed (Participants) | 94 | 100
  Pain affect normal work last 24hrs-visit8 | 5.0 (3.1) | 5.5 (3.2)
  Pain affect relation with others last 24hrs-visit2 | 3.8 (2.8) | 4.1 (3.0)
  Pain affect relation with others last 24hrs-visit5: number analyzed (Participants) | 101 | 102
  Pain affect relation with others last 24hrs-visit5 | 3.5 (2.7) | 3.5 (2.6)
  Pain affect relation with others last 24hrs-visit6: number analyzed (Participants) | 95 | 99
  Pain affect relation with others last 24hrs-visit6 | 3.2 (2.6) | 3.6 (2.7)
  Pain affect relation with others last 24hrs-visit7: number analyzed (Participants) | 88 | 96
  Pain affect relation with others last 24hrs-visit7 | 3.2 (2.7) | 3.6 (2.7)
  Pain affect relation with others last 24hrs-visit8: number analyzed (Participants) | 94 | 100
  Pain affect relation with others last 24hrs-visit8 | 3.4 (2.6) | 4.0 (2.8)
  Pain affect sleep last 24hrs-visit2 | 5.0 (2.9) | 5.1 (2.9)
  Pain affect sleep last 24hrs-visit5: number analyzed (Participants) | 101 | 102
  Pain affect sleep last 24hrs-visit5 | 4.3 (2.7) | 4.1 (2.8)
  Pain affect sleep last 24hrs-visit6: number analyzed (Participants) | 95 | 99
  Pain affect sleep last 24hrs-visit6 | 3.8 (2.5) | 3.9 (2.5)
  Pain affect sleep last 24hrs-visit7: number analyzed (Participants) | 88 | 96
  Pain affect sleep last 24hrs-visit7 | 3.8 (2.6) | 3.9 (2.7)
  Pain affect sleep last 24hrs-visit8: number analyzed (Participants) | 94 | 100
  Pain affect sleep last 24hrs-visit8 | 3.8 (2.6) | 4.1 (2.8)
  Pain affect enjoyment of life last 24hrs-visit2 | 5.3 (3.2) | 5.7 (3.1)
  Pain affect enjoyment of life last 24hrs-visit5: number analyzed (Participants) | 101 | 102
  Pain affect enjoyment of life last 24hrs-visit5 | 4.6 (3.0) | 4.6 (2.8)
  Pain affect enjoyment of life last 24hrs-visit6: number analyzed (Participants) | 95 | 99
  Pain affect enjoyment of life last 24hrs-visit6 | 4.4 (3.0) | 4.7 (3.0)
  Pain affect enjoyment of life last 24hrs-visit7: number analyzed (Participants) | 88 | 96
  Pain affect enjoyment of life last 24hrs-visit7 | 4.0 (2.8) | 4.8 (3.1)
  Pain affect enjoyment of life last 24hrs-visit8: number analyzed (Participants) | 94 | 100
  Pain affect enjoyment of life last 24hrs-visit8 | 4.6 (2.9) | 4.9 (3.1)
  Mean of seven interference items-visit2 | 5.0 (2.3) | 5.4 (2.4)
  Mean of seven interference items-visit5: number analyzed (Participants) | 101 | 102
  Mean of seven interference items-visit5 | 4.4 (2.2) | 4.4 (2.3)
  Mean of seven interference items-visit6: number analyzed (Participants) | 95 | 99
  Mean of seven interference items-visit6 | 4.1 (2.2) | 4.5 (2.4)
  Mean of seven interference items-visit7: number analyzed (Participants) | 88 | 96
  Mean of seven interference items-visit7 | 4.0 (2.2) | 4.5 (2.5)
  Mean of seven interference items-visit8: number analyzed (Participants) | 94 | 100
  Mean of seven interference items-visit8 | 4.3 (2.4) | 4.7 (2.7)

8. Secondary Outcome: The Change of Bowel Movement by Visit
Description: Number pf bowel movements(BM) and number of days the subjects had a bowel movement in the last 7 days before the study visit will be summarized at visit2(day0) ,visit5(day7),visit6(day14),visit7(day21), visit8(day28)..
Time Frame: visit2 (day 0) to visit8 (week 4 or early discontinue/withdrawal from study)
Population: FAP
Measure: Mean (Standard Deviation); unit: Bowel movement/day
Arm/Group | Oxycodone/Naloxone | Oxycodone
Number analyzed (Participants) | 107 | 106
Bowel movement/day
  Number of BM baseline in last 7 days-visit2 | 2.9 (1.7) | 3.1 (1.7)
  Number of BM baseline in last 7 days-visit5: number analyzed (Participants) | 101 | 102
  Number of BM baseline in last 7 days-visit5 | 3.7 (2.5) | 3.5 (2.6)
  Number of BM baseline in last 7 days-visit6: number analyzed (Participants) | 95 | 99
  Number of BM baseline in last 7 days-visit6 | 4.2 (3.4) | 3.9 (2.3)
  Number of BM baseline in last 7 days-visit7: number analyzed (Participants) | 88 | 96
  Number of BM baseline in last 7 days-visit7 | 4.2 (2.8) | 3.9 (2.3)
  Number of BM baseline in last 7 days-visit8: number analyzed (Participants) | 97 | 101
  Number of BM baseline in last 7 days-visit8 | 3.7 (2.5) | 3.5 (2.6)
  Number of days with BM in last 7 days-visit2 | 2.8 (1.5) | 3.0 (1.6)
  Number of days with BM in last 7 days-visit5: number analyzed (Participants) | 101 | 102
  Number of days with BM in last 7 days-visit5 | 3.1 (1.7) | 3.0 (1.6)
  Number of days with BM in last 7 days-visit6: number analyzed (Participants) | 95 | 99
  Number of days with BM in last 7 days-visit6 | 3.4 (1.6) | 3.5 (1.7)
  Number of days with BM in last 7 days-visit7: number analyzed (Participants) | 88 | 96
  Number of days with BM in last 7 days-visit7 | 3.6 (1.7) | 3.5 (1.8)
  Number of days with BM in last 7 days-visit8: number analyzed (Participants) | 97 | 101
  Number of days with BM in last 7 days-visit8 | 3.3 (1.8) | 3.2 (1.9)

9. Secondary Outcome: The Chage of Symptoms of Constipation Based on Laxative Use From visit5 to visit8
Description: At Visit5(day7) and visit8(day28) number of bisacodyl taken(Number of laxative tablets took during the last 7 days (per week) and Daily number of laxative tablets took during the last 7 days (per day)*) for OXN PR and OXY PR groups
Time Frame: visit 5 taking place at week 1 to visit8 taking place at week 4 or early discontinue/withdrawal from study where applicable
Population: FAP
Measure: Mean (Standard Deviation); unit: laxatives/day
Arm/Group | Oxycodone/Naloxone | Oxycodone
Number analyzed (Participants) | 107 | 106
laxatives/day
  Daily number of bisacodyl taken at Visit5 | 0.9 (0.9) | 1.1 (0.9)
  Daily number of bisacodyl taken at Visit8 | 0.9 (0.9) | 0.9 (0.9)

ADVERSE EVENTS:
Time Frame: The adverse event data were collected from 2013 Jun to 2014 Aug, which is about 14 months. The time frame of AE collection for each subject is about 6 weeks.
Description: same as clinicaltrials.gov definition
Arm/Group | Oxycodone/Naloxone | Oxycodone
All-Cause Mortality (participants affected / at risk) | 8/114 | 4/111
Serious Adverse Events (participants affected / at risk) | 14/114 | 12/111
Other Adverse Events (participants affected / at risk) | 72/114 | 76/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone/Naloxone (N=114) | Oxycodone (N=111)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bone marrow failure (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intentional overdose* (Social circumstances) | 0 (0) | 1 (1) — SAEs in Subject 080806 reported as 2 PT's: Intentional overdose and Suicide attempt and were calculated as 2 SAEs.
Intra-abdominal hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Suicide attempt (Social circumstances) | 0 (0) | 1 (1) — SAEs in Subject 080806 reported as 2 PT's: Intentional overdose and Suicide attempt and were calculated as 2 SAEs.
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone/Naloxone (N=114) | Oxycodone (N=111)
Vomiting (Gastrointestinal disorders) | 27 (63) | 22 (57)
Abdominal distension (Gastrointestinal disorders) | 6 (17) | 6 (17)
Nausea (Gastrointestinal disorders) | 9 (13) | 12 (19)
Pyrexia (General disorders) | 6 (8) | 6 (13)
Abdominal pain upper (General disorders) | 1 (14) | 2 (5)
Fatigue (General disorders) | 4 (4) | 9 (11)
Decreased appetite (General disorders) | 2 (3) | 10 (10)
Dizziness (General disorders) | 3 (3) | 6 (8)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 6 (8)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 4 (4)
Urinary tract infection (Renal and urinary disorders) | 4 (4) | 5 (5)
Constipation (Gastrointestinal disorders) | 0 (0) | 6 (8)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Bone marrow failure (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3)
Hyperhidrosis (General disorders) | 2 (2) | 4 (4)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 1 (1)
GGT increased (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Somnolence (General disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-03-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT01885182/Prot_000.pdf
  • Statistical Analysis Plan (2014-12-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT01885182/SAP_001.pdf